CLINICAL TRIAL: NCT06578936
Title: The Effect of Abdominal Massage and Warm Application on Excretory Activity in Patients Undergoing Total Knee Replacement With Spinal Anesthesia
Acronym: Abdominal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe Demirtaş (Other)
Responsible Party: Sponsor-Investigator, Ayşe Demirtaş, student researcher, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MU-DEMIRTAS-01
Record Dates: First submitted 2024-08-09; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Total Knee Replacement
Keywords: heat application; constipation; intestinal motility; spinal anesthesia
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: A prospective, parallel, two-arm, randomized controlled clinical trial
Who Masked: Participant
Masking Description: A biostatistician who is not involved in the study will be randomly assigned to groups A and B, which are formed by a biostatistician in the computer environment. As a result of the draw of lots, whether group A and B will be the study or control group will be determined by a coin toss at the beginning of the study. The information showing that the patients included in the research sample are assigned to groups A and B according to the randomization table will be placed in an opaque envelope. This envelope will be kept by the coordinator researcher (GAU), and when the researcher (AD) goes to the patient for the application, he/she will open the envelope after filling out the "Informed Consent Form" and learn which group the patient is in
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- abdominal massage and warm application group (Experimental): The experimental group will receive abdominal massage and warm application 2 times a day, morning and evening, until defecation, starting from the evening of the first day after the surgical intervention.
  Interventions: Other: abdominal massage andwarm application
- control group (No Intervention): In the control group, bowel sounds will be listened during hot application and abdominal massage hours, daily laxative use will be determined and recorded in the Excretory Activity Form.

INTERVENTIONS:
Other: abdominal massage andwarm application — Abdominal massage and hot application will be applied to the patients at least 30 minutes after the morning and evening meals (08:30 am, 20:30 pm) for 15 minutes each, similar to the literature. The hot application will be applied to the abdominal area with a hot water thermophore for 15 minutes before the abdominal massage. After the hot application, abdominal massage will be started. In the abdominal massage, which will be applied clockwise to stimulate bowel movements, four basic movements will be used: superficial exertion, deep exertion, petrisage and vibration.
  Arms: abdominal massage and warm application group

SUMMARY:
The aim of this study was to determine the effect of abdominal massage and warm application on the excretory activity (time of first bowel sounds, defecation time and the amount of laxative used until discharge) after total knee replacement surgery performed with spinal anesthesia.

DETAILED DESCRIPTION:
Abdominal massage and hot application will be applied to the patients at least 30 minutes after the morning and evening meals (08:30 am, 20:30 pm) for 15 minutes each, similar to the literature. The hot application will be applied to the abdominal area with a hot water thermophore for 15 minutes before the abdominal massage. After the hot application, abdominal massage will be started. In the abdominal massage, which will be applied clockwise to stimulate bowel movements, four basic movements will be used: superficial exertion, deep exertion, petrisage and vibration. Abdominal massage will be applied to the patients in accordance with the Abdominal Massage Application Checklist created by the researcher in line with the literature.

Warm application and abdominal massage will be applied to the study group from the first evening of the total knee replacement procedure, and the application will continue in the morning and evening hours until the first defecation. After the application, bowel sounds will be listened to in accordance with the application steps. In the control group, bowel sounds will be listened to at times corresponding to the hours of hot application and abdominal massage, daily laxative use will be determined and recorded in the Excretory Activity Form.

ELIGIBILITY:
Inclusion Criteria:

* Written and verbal permission was obtained to participate in the study,
* 18 years of age or older,
* Conscious, oriented and cooperative,
* Speaks and understands Turkish,
* Total knee replacement with spinal anesthesia planned,
* No condition in which abdominal massage is contraindicated (inflammatory bowel disease, presence of abdominal tumors, surgical intervention or radiotherapy to the abdominal area, presence or suspicion of ileus, and pregnancy),
* No physician-diagnosed chronic constipation,
* Mobilized,
* Patients who do not have problems with transition to oral feeding and can be fed orally will be included.

Exclusion Criteria:

* Written and verbal permission to participate in the research could not be obtained,
* Under 18 years of age,
* Unconscious, disoriented and uncooperative,
* Can speak Turkish but cannot understand it,
* Total knee replacement with general anesthesia planned,
* Any condition in which abdominal massage is contraindicated (inflammatory bowel disease, presence of abdominal tumors, surgical intervention or radiotherapy to the abdominal area, presence or suspicion of ileus, and pregnancy),
* Physician-diagnosed chronic constipation,
* Non-mobilized,
* Patients who have problems with transition to oral feeding and who cannot be fed orally will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
time for bowel sounds to return | 1-3.days
  The time of return of bowel sounds in the morning and evening will be assessed and recorded on the Excretory Activities Form.
time to defecate | 1-3.day
  the effect of abdominal massage and warm application on defecation time after total knee replacement

SECONDARY OUTCOMES:
risk of constipation | 1-3.days
  postoperative defecation status will be recorded on the excretory activity form and the risk of constipation will be assessed
laxative use | 1-3.days
  The amount of medication used to facilitate defecation is assessed in the morning and evening and recorded on the Excretory Activities Form.

CONTACTS AND LOCATIONS:
Overall Officials: gülay altun uğraş, PhD, Study Director — mersin univercity
Locations (2):
- Turkey (Türkiye) (2):
  - Adana city hospital, Adana
  - Mersin Univercity, Mersin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Axelby E, Kurmis AP. Gabapentoids in knee replacement surgery: contemporary, multi-modal, peri-operative analgesia. J Orthop. 2019 Jul 2;17:150-154. doi: 10.1016/j.jor.2019.06.031. eCollection 2020 Jan-Feb. PMID 31879495
- [Result] Jaber A, Hemmer S, Klotz R, Ferbert T, Hensel C, Eisner C, Ryang YM, Obid P, Friedrich K, Pepke W, Akbar M. Bowel dysfunction after elective spinal surgery: etiology, diagnostics and management based on the medical literature and experience in a university hospital. Orthopade. 2021 Jun;50(6):425-434. doi: 10.1007/s00132-020-04034-z. PMID 33185695
- [Result] Aydinli A, Karadag S. "Effects of abdominal massage applied with ginger and lavender oil for elderly with constipation: A randomized controlled trial". Explore (NY). 2023 Jan-Feb;19(1):115-120. doi: 10.1016/j.explore.2022.08.010. Epub 2022 Aug 20. PMID 36058824
- [Result] Nagashima Y, Oda H, Igaki M, Suzuki M, Suzuki A, Yada Y, Tsuchiya S, Suzuki T, Ohishi S. Application of heat- and steam-generating sheets to the lumbar or abdominal region affects autonomic nerve activity. Auton Neurosci. 2006 Jun 30;126-127:68-71. doi: 10.1016/j.autneu.2006.02.002. Epub 2006 Mar 6. PMID 16624632